CLINICAL TRIAL: NCT02804139
Title: Physical Therapy in Addition to Standard Care Following C-Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jennifer Y Stone, Supervisor, Clinical Rehabilitation Services, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003233
Record Dates: First submitted 2016-05-10; First posted 2016-06-17 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Low Back Pain; Pelvic Pain; Scar Tissue; Adhesions
Keywords: Cesarean Section; Postpartum issues
MeSH Terms: conditions — Low Back Pain; Pelvic Pain; Cicatrix; Tissue Adhesions | interventions — Standard of Care; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (Active Comparator): Standard Care after C-section with no additional physical therapy.
  Interventions: Other: Standard Care
- Standard care plus physical therapy (Experimental): Subjects attend 1 to 2 physical therapy sessions per week for 6 weeks beginning 8-10 weeks post-C section. The physical therapy program includes scar management, core retraining, and lumbar and pelvic joint mobilization
  Interventions: Other: Standard care plus physical therapy

INTERVENTIONS:
Other: Standard care plus physical therapy — Subjects attend 1 to 2 physical therapy sessions per week for 6 weeks beginning 8-10 weeks post-C section. The physical therapy program includes scar management, core retraining, and lumbar and pelvic joint mobilization.
  Arms: Standard care plus physical therapy
Other: Standard Care — Standard Care after C-section with no additional physical therapy.
  Arms: Standard care

SUMMARY:
The purpose of this study is to determine whether a physical therapy program which includes scar management, core retraining, and lumbar and pelvic joint mobilization will significantly impact the postpartum recovery following Cesarean section during the immediate postpartum period and during the first 1.5 years following childbirth.

All patients who enroll in the study will receive standard treatment following a C-section delivery. Subjects will be randomized into one of two groups; one group will receive physical therapy in addition to standard post C-section treatment, and the other group will receive standard post C-section treatment with no additional physical therapy. Both groups will complete questionnaires regarding their pain and recovery from C-section delivery to determine if there is a difference in recovery between the group receiving physical therapy and the group not receiving physical therapy.

DETAILED DESCRIPTION:
Cesarean section (C-section) represents the most commonly performed inpatient surgical procedure, with recent prevalence estimates of 1.3 million annually (approximately 22% of first births) in the United States. Currently, postoperative recovery support is typically characterized by verbal and written instructions regarding lifting and pelvic rest as well as slow return to activity and exercise.

There are multiple known complications during and after the postpartum period following Cesarean section deliveries. Some of the most common are back pain (up to 53% prevalence reported), bowel and bladder issues (20-30% prevalence reported), and scar tissue/adhesions. Multiple studies have indicated a higher incidence of low back and pelvic girdle pain in patients following Cesarean section compared to an unassisted vaginal delivery (estimates range from 2-5 times increase).

The purpose of this study is to determine whether a physical therapy program which includes scar management, core retraining, and lumbar and pelvic joint mobilization will significantly impact the postpartum recovery following Cesarean section during the immediate postpartum period and during the first 1.5 years following childbirth.

ELIGIBILITY:
Inclusion Criteria:

* Caesarean section delivery, English speaking

Exclusion Criteria:

* Heart problems, postpartum eclampsia, any medical issue which contraindicates exercise, active untreated infection, chronic narcotic use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index | 8 weeks, 14 weeks, 6 months, 1 year, and 1.5 years after C-section
  The change in the Oswestry Disability Index from 8 week baseline to subsequent time points.

SECONDARY OUTCOMES:
Change in Visual Analogue Pain Scale Rating. | 8 weeks, 14 weeks, 6 months, 1 year, and 1.5 years after C-section
  The change in visual analogue pain scale ratings from 8 week baseline to subsequent time points for the neck, shoulders, low back, pelvis / hips, lower legs and "other" body area

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stone, PT, DPT, OCS, Principal Investigator — University of Missouri Health Care
Locations (1):
- University of Missouri Health Care, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No